CLINICAL TRIAL: NCT00364442
Title: A Repeat Dose, Randomised, Double Blind, 2-way Crossover Study to Assess the Safety and Systemic Exposure of an Investigational Formulation Compared to Concurrent Administration of Individual Fluticasone Propionate 50 and Salmeterol 50 DISKUS Inhalers in Subjects Aged 18 - 55 Years With Mild Asthma
Brief Title: Repeat Dose Study of Fluticasone Propionate/Salmeterol Versus Fluticasone Propionate + Salmeterol In Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SAS10019
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): investigational drug
  Interventions: Drug: fluticasone propionate/salmeterol

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol — investigational drug

SUMMARY:
A new formulation of Fluticasone propionate/Salmeterol comparing a lower dose of fluticasone propionate and salmeterol was compared with concurrent administration of fluticasone propionate and salmeterol. Administration occurred over 14 days and tolerability, PK (pharmacokinetic) and PD (pharmacodynamic) measurements were performed.

ELIGIBILITY:
Inclusion criteria:

* Documented history of mild or intermittent asthma
* Have PEF and FEV1>80% predicted
* Not a smoker
* BMI of 19 - 29

Exclusion criteria:

* Have had a life threatening episode of asthma
* Have had a respiratory tract infection in the last four weeks
* Have other respiratory disease
* Have taken certain medications within restricted time periods

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01-28 (Actual); Primary Completion 2005-04-13 (Actual); Study Completion 2005-04-13 (Actual)

PRIMARY OUTCOMES:
The primary objective was to look at the safety and tolerability of a low dose of fluticasone propionate/salmeterol compared to concurrent administration of fluticasone propionate and salmeterol | Administration occurred over 14 days and tolerability

SECONDARY OUTCOMES:
Comparing changes in PD parameters & PK parameters between a low dose of fluticasone propionate/salmeterol compared to concurrent administration of fluticasone propionate and salmeterol | Administration occurred over 14 days and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study SAS10019 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/SAS10019?search=study&search_terms=SAS10019#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAS10019 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register